CLINICAL TRIAL: NCT07158918
Title: A Multicenter, Open-label, Phase 1b/2 Trial of ABL103, a Bispecific Antibody of B7-H4 and 4-1BB, in Combination With Pembrolizumab With/Without Taxane in Subjects With Selected, Progressive, Locally Advanced (Unresectable) or Metastatic Solid Tumors
Brief Title: ABL103 in Combination With Pembrolizumab, With or Without Taxane in Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ABL Bio, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABL103-1002; KEYNOTE-G16 (Other: Merck Sharp & Dohme LLC); MK-3475-G16 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2025-08-08; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — pembrolizumab; taxane

STUDY DESIGN:
Intervention Model Description: Dose escalation and Dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ABL103 (DL1) + pembrolizumab (Experimental): Safety Lead-in Part 1
  Interventions: Drug: ABL103; Drug: KEYTRUDA® (pembrolizumab)
- ABL103 (DL2-1) + pembrolizumab + taxane (Experimental): Safety Lead-in Part 2
  Interventions: Drug: ABL103; Drug: KEYTRUDA® (pembrolizumab); Drug: Taxane
- ABL103 (DL2) + pembrolizumab + taxane (Experimental): Safety Lead-in Part 2
  Interventions: Drug: ABL103; Drug: KEYTRUDA® (pembrolizumab); Drug: Taxane
- Group 1) ABL103 + pembrolizumab + taxane (Experimental): Dose-expansion Part
  Interventions: Drug: ABL103; Drug: KEYTRUDA® (pembrolizumab); Drug: Taxane
- Group 2) ABL103 + pembrolizumab + taxane (Experimental): Dose-expansion Part
  Interventions: Drug: ABL103; Drug: KEYTRUDA® (pembrolizumab); Drug: Taxane

INTERVENTIONS:
Drug: ABL103 — IV infusion
Drug: KEYTRUDA® (pembrolizumab) — IV infusion
Drug: Taxane — IV infusion
  Arms: ABL103 (DL2) + pembrolizumab + taxane; ABL103 (DL2-1) + pembrolizumab + taxane; Group 1) ABL103 + pembrolizumab + taxane; Group 2) ABL103 + pembrolizumab + taxane

SUMMARY:
This study is to assess the safety and antitumor activity of ABL103 plus pembrolizumab, with or without taxane, in advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject must understand and be willing to provide informed consent and be able to comply with the study procedures and restrictions.
* Subjects must be ≥18 years of age on the day of signing the informed consent form (ICF).
* Subject must have a histologically or cytologically confirmed locally advanced unresectable, or metastatic solid tumor.
* Subject must be relapsed or be refractory to available standard therapy or they must be intolerant of available standard therapy.
* Subject must meet Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 assessed 7 days before the first administration of the study drug.
* Subjects must be recovered from AEs from prior therapy to Grade 1 or the baseline grade more than 14 days prior to the first administration of the study drug, except alopecia or Grade 2 toxicities that are deemed stable or irreversible (e.g., peripheral neuropathy)
* Subjects who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Subject with endocrine-related AEs who are adequately treated with hormone replacement or subjects who have ≤Grade 2 neuropathy are eligible.
* Subjects must have adequate hematologic, renal, hepatic, and thyroid function at screening and within 7 days prior to the first administration of study drug.
* Female subjects who are not surgically sterile or postmenopausal must agree to use a highly effective method of birth control (2 methods strongly recommended) during the study and for 6 months following the last dose of ABL103/pembrolizumab.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening and within 7 days prior to Cycle 1 Day 1 (C1D1).
* Male subjects with female partner(s) of childbearing potential must agree to use contraception and and must not donate sperm during the treatment period with ABL103 and taxane and for at least 6 months after the final administration of ABL103 and taxane.
* Male subjects with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom throughout the study period, and for at least 6 months after the final administration of ABL103 and taxane, and during the partner's pregnancy or breastfeeding period. When using a male condom, the partner must also use an additional method of contraception acceptable for female subjects.

Exclusion Criteria:

* Subject has received prior anticancer monoclonal antibody treatment or investigational therapy (agent or device) for which the pharmacologic or toxicity profile is not expected to have resolved prior to the first administration of the study drug. A minimum of 28 days is generally recommended for agents with known delayed toxicities or prolonged biological activity, unless otherwise justified.
* Subject has received prior radiotherapy within 2 weeks of the first administration of study drug, or has radiation-related toxicities, requiring corticosteroids.
* Subject has received any prior immunotherapy and was discontinued from the treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
* Subject has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study treatment.
* Subject has risk factors for bowel obstruction or bowel perforation, including, but not limited to a history of acute diverticulitis, intra-abdominal abscess, and abdominal carcinomatosis. Subjects with ovarian cancer with a history of abdominal carcinomatosis can be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | Day 1 to Day 21 (Safety Lead-in Part 1) and Day 1 to Day 28 (Safety Lead-in Part 2)
Incidence of Treatment-Emergent Adverse Events (TEAEs), Treatment-Related AEs, Serious AEs (SAEs), and Infusion-Related Reactions (IRRs) | From baseline through study completion, an average of 12 months
Recommended Dose for Expansion (RDE) Determination | From baseline through study completion, an average of 12 months
Objective Response Rate (ORR) | Up to approximately 30 months
Disease Control Rate (DCR) | Up to approximately 30 months

SECONDARY OUTCOMES:
Preliminary Objective Response Rate (ORR) | Up to approximately 30 months
Preliminary Disease Control Rate (DCR) | Up to approximately 30 months
Incidence of Anti-Drug Antibodies (ADA) | From baseline through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sangmi Lee, Study Director — ABL Bio
Locations (6):
- UH Cleveland Medical Center, Cleveland, Ohio, United States
- PASO Medical, Frankston, Victoria, Australia
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided